CLINICAL TRIAL: NCT05838937
Title: The Usefulness of Myocardial Work IndeX in ExtraCorporeal Membrane Oxygenation Patients
Acronym: MIX-ECMO
Status: Not yet recruiting | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: I.Medizinische Klinik, Universitätsklinikum Mannheim (Unknown); University Hospital, Limoges (Other)
Responsible Party: Principal Investigator, Balint Karoly Lakatos, Assistant Professor, Semmelweis University Heart and Vascular Center
Other Study IDs: BMEÜ/4229- 1 /2022/EKU
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Echocardiography; Mechanical Circulatory Support; Myocardial Failure; Cardiogenic Shock; Extracorporeal Membrane Oxygenation Complication
Keywords: Echocardiography; Myocardial work index; Cardiogenic shock; Extracorporeal Membrane Oxygenation Therapy
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Investigation cohort: Cardiogenic shock patients from any cause receiving veno-arterial extracorporeal membrane oxygenation

SUMMARY:
Investigation of the potential prognostic role of non-invasive myocardial work in patients receiving veno-arterial extracorporeal membrane oxygenation therapy.

DETAILED DESCRIPTION:
The study aims to examine the prognostic role of non-invasive myocardial work in veno-arterial extracorporeal membrane oxygenation therapy patients. Subjects with cardiogenic shock regardless of etiology will be enrolled 48-72 hours after the initiation of mechanical circulatory support. It is hypothesized that non-invasive myocardial work may be an independent prognosticator of the outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older age
* Severe cardiogenic shock requiring the initiation of VA-ECMO therapy
* Stabile hemodynamic state and oxigenation with VA-ECMO and vasoactive support
* Informed written consent (due to the nature of the study, from a legally eligible relative of the patient)

Exclusion Criteria:

* Younger than 18 years of age
* Unstable hemodynamic state or suboptimal oxigenation despite established VA-ECMO and vasoactive support
* Severe neurological damage or confirmed brain death at the time of enrollment which squarely indicates therapy limitation and poor short-term outcome
* Transesophageal echocardiography is contraindicated
* Suboptimal echocardiographic window

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Altogether 100 cardiogenic shock patients receiving veno-arterial extracorporeal membrane oxygenation therapy will be enrolled regardless the etiology. Both peripherially and centrally cannulated patients are eligible. Considering that the two populations are typically quite different in terms of indication for the therapy (ACS- or decompensated chronic heart failure-associated CS vs. cardiac surgery population), a balanced enrollment of the two methods will be facilitated. All LV venting options are eligible for enrollment, however, if utilized, the mode of LV unloading (central left atrial vent, Impella, transaortic LV pigtail catheter etc.) will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality, need for long-term mechanical circulatory support or heart transplantation | 30 days
  The total number of patients who die from cardiovascular cause, or require for transition to long-term mechanical circulatory support (LVAD/BiVAD), or heart transplantation

SECONDARY OUTCOMES:
All-cause mortality | 30 days
  Death from any cause during the study period
Need for renal replacement therapy | 30 days
  The total number of patients who need for renal replacement therapy during intensive care
Successful weaning from mechanical ventilation | 30 days
  The total number of patients who can be successfully weaned from invasive mechanical ventilation
Discharge from intensive care unit | 30 days
  The total number of patients who are discharged from intensive care unit
Discharge from hospital | 30 days
  The total number of patients who are discharged from hospital
Ventilator-free days | 30 days
  Days spent without invasive mechanical ventilation
VA-ECMO-free days | 30 days
  Days spent without VA-ECMO support

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, BP, Hungary

IPD SHARING:
Plan to Share IPD: Undecided